CLINICAL TRIAL: NCT00893061
Title: A Prospective, Randomized, Open-label, Multicenter Study Evaluating the Effects on Cognitive Functions of Adjuvant Endocrine Therapy in Postmenopausal Women With Breast Cancer.
Brief Title: Letrozole, Anastrozole, Exemestane, or Tamoxifen Citrate in Treating Postmenopausal Women With Breast Cancer
Acronym: MNEMOSYNE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MNEMOSYNE-0712; 2008-003620-32 (EudraCT Number)
Record Dates: First submitted 2009-05-02; First posted 2009-05-05 (Estimated); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer
Keywords: stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; estrogen receptor-positive breast cancer; progesterone receptor-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; exemestane; Letrozole; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Experimental): Patients receive oral tamoxifen citrate once daily for 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: tamoxifen citrate
- Arm II (Experimental): Patients receive an oral aromatase inhibitor (letrozole, anastrozole, or exemestane) once daily for 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: anastrozole; Drug: exemestane; Drug: letrozole

INTERVENTIONS:
Drug: anastrozole — Given orally
  Arms: Arm II
Drug: exemestane — Given orally
  Arms: Arm II
Drug: letrozole — Given orally
  Arms: Arm II
Drug: tamoxifen citrate — Given orally
  Arms: Arm I

SUMMARY:
RATIONALE: Estrogen can cause the growth of breast cancer cells. Aromatase inhibitors, such as letrozole, anastrozole, and exemestane, may fight breast cancer by lowering the amount of estrogen the body makes. Hormone therapy, using tamoxifen citrate, may fight breast cancer by blocking the use of estrogen by the tumor cells. It is not yet known whether aromatase inhibitors or tamoxifen citrate have less effect on memory in patients receiving treatment for breast cancer.

PURPOSE: This randomized phase III trial is studying letrozole, anastrozole, or exemestane to see how they effect memory compared with tamoxifen citrate in treating postmenopausal women with breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate verbal episodic memory in patients with breast cancer after 6 months of treatment with aromatase inhibitors (AI) vs tamoxifen citrate.

Secondary

* To evaluate cognitive functions of these patients at month 6 and 12 of treatment.
* To evaluate the psychological and social impact on these patients at month 6 and 12 of treatment.

OUTLINE: This is a multicenter study.

Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral tamoxifen citrate once daily for 1 year in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive an oral aromatase inhibitor (letrozole, anastrozole, or exemestane) once daily for 1 year in the absence of disease progression or unacceptable toxicity.

Patients undergo cognitive, psychological, social, and quality of life assessments every 6 months using the CDS scale, the Edinburgh Handedness Inventory, the Mini Mental Test, the French version of the National Adult Reading Test, the Benton Visual Retention test, the direct and indirect capacities of the WAIS-R, the WMS sequential visual-spatial capacity, the dual task test, categorical and formal verbal fluency, the Trail making test, the Stroop test, the Wisconsin Card Sorting test, the choice reaction time test, the sequential visual spatial capacity, the HADS scale, IADL, and QLQ-C30 questionnaires.

After completion of study treatment, patients are followed for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer
* No metastatic disease
* Meets criteria for initiating adjuvant endocrine therapy
* Hormone receptor status:

  * Estrogen receptor- and/or progesterone receptor-positive disease

PATIENT CHARACTERISTICS:

* Postmenopausal, defined as no menstruation for ≥ 1 year, confirmed by a measurement of FSH and 17-beta-estradiol
* Karnofsky performance status 80-100%
* Native speaker of French
* Beneficiary of a French Social Security insurance plan
* No prior cognitive disorders
* No depression or other confirmed active psychiatric disease
* Able to undergo the medical monitoring of the trial due to geographic, social or psychological reasons
* No personal or family history of thromboembolic disease

PRIOR CONCURRENT THERAPY:

* No prior adjuvant chemotherapy
* No concurrent follow-up participation on another study
* No concurrent treatment with psychotropic substances (i.e., long half life benzodiazepines, antipsychotics, anticholinesterase)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-03-16 (Actual); Primary Completion 2012-04-04 (Actual); Study Completion 2014-11-26 (Actual)

PRIMARY OUTCOMES:
Changes in verbal episodic memory performance after 6 months of treatment, using the Rey Auditory Verbal Learning Test | From baseline to 6 months of treatment

SECONDARY OUTCOMES:
Changes in other cognitive functions at 6 and 12 months of treatment | From baseline to 6 and 12 months of treatment
Psychological and social impact at 6 and 12 months of treatment, using the HADS scale and quality of life questionnaires (i.e., IADL and QLQ-C30) | From baseline to 6 and 12 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Le Rhun, Principal Investigator — Centre Oscar Lambret
Locations (3):
- France (3):
  - Centre Oscar Lambret, Lille
  - Centre Eugene Marquis, Rennes
  - Centre Paul Strauss, Strasbourg